CLINICAL TRIAL: NCT00194506
Title: Cyber Disease Management: Using the World Wide Web to Share the Medical Record With Patients at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Center for Health Management Research (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 00-3882-E/A 05
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-04-14 (Estimated); Status verified 2006-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Health Education; Information Technology; Disease Management; Internet; Patient Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Health Education

INTERVENTIONS:
Behavioral: Internet co-management module

SUMMARY:
This is a 12-month randomized, controlled trial of a Web-based diabetes co-management module among type 2 patients at the University of Washington's Roosevelt General Internal Medicine Clinic.

DETAILED DESCRIPTION:
We will conduct a randomized controlled trial to determine whether a fully computerized, diabetes mellitus (DM) disease-management module (known as Cyber-DM) can improve the quality of adult diabetes care. The module will be Web-based, include a graphical HTML "front end" user interface, and will be incorporated into each patient's existing Web-based electronic medical record --the Medical Information Networked Database (MIND) repository at the University of Washington Academic Medical Centers. This Web site will include five components that will enable patients to interact asynchronously from their homes with their clinic-based providers:

1. An integrated view of their actual medical record as it relates to diabetes care that can generate customized patient education materials.
2. Real-time clinical reminders of the need to obtain preventive services such as HbA1c, urine-protein and cholesterol determinations, and retinal examinations.
3. An electronic version of the SDMTM diabetes-care algorithms indicating where on the "road-map" to adequate control they currently stand treatment-wise.
4. The ability to download glucometer readings and medication-use information from home directly into the MIND repository.
5. Secure email communication between patients, their primary care physicians, and clinic staff.

A total of 80-85 diabetic patients who are regular utilizers of the UW's General Internal Medicine Clinic and who have home Internet access will be randomized to the experimental and control arms of the trial. Control subjects will receive usual care. We hypothesize that use of Cyber-DM will increase compliance with guideline-indicated care processes, improve glycemic control, and reduce utilization costs. A trial this size would have the statistical power to detect a change in HbA1c of 0.50%. Secure Socket Layer technology, session specific "cookie" files, and a custom database application that manages logins/passwords and audits all accesses to the system will provide security for this information tool.

ELIGIBILITY:
Inclusion Criteria:

* computer and Internet access at home
* receiving care for type 2 diabetes at the University of Washington, General Internal Medicine Clinic, Roosevelt

Exclusion Criteria:

* non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 2002-08; Study Completion 2006-05

PRIMARY OUTCOMES:
Hemoglobin A1c

SECONDARY OUTCOMES:
Utilization

CONTACTS AND LOCATIONS:
Overall Officials: Harold I. Goldberg, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, General Internal Medicine Clinic, Roosevelt, Seattle, Washington, United States

REFERENCES:
- [Derived] Ralston JD, Hirsch IB, Hoath J, Mullen M, Cheadle A, Goldberg HI. Web-based collaborative care for type 2 diabetes: a pilot randomized trial. Diabetes Care. 2009 Feb;32(2):234-9. doi: 10.2337/dc08-1220. Epub 2008 Nov 18. PMID 19017773